CLINICAL TRIAL: NCT03552107
Title: Real World Experience With Lorcaserin for Weight Management
Brief Title: Lorcaserin: Real World Experience in an Insurance-Based Weight Management Clinic
Status: Completed | Type: Observational
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corporate Vice President, Scripps Whittier Diabetes Institute
Other Study IDs: Lorcaserin
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Weight Loss; Overweight
Keywords: Lorcaserin; Belviq
MeSH Terms: conditions — Obesity; Weight Loss; Overweight | interventions — lorcaserin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Group - Lorcaserin Treated: The group in this study will be all patients who initiated therapy with Lorcaserin during the review period.
  Interventions: Drug: Lorcaserin

INTERVENTIONS:
Drug: Lorcaserin — Treatment initiation with Lorcaserin
  Other Names: Belviq

SUMMARY:
This is a retrospective, descriptive study that involves de-identified data consisting of weight changes, pertinent vital signs and laboratory values influenced by body weight, and healthcare utilization of patients prescribed lorcaserin at The Center for Weight Management at the Scripps Clinic in San Diego, CA.

DETAILED DESCRIPTION:
All patients who initiated treatment with Lorcaserin during the review period will undergo chart review. The primary endpoint will be weight change in patients on Lorcaserin and average duration of Lorcaserin treatment over time (up to 1 year). Secondary endpoints will include changes in vital signs, liver function, glucose, and lipids. In addition, time on treatment, reasons for discontinuation of medication, and changes in healthcare utilization (to include inpatient and outpatient utilization) will be examined. This is a retrospective, one-arm observational study that will include chart reviews of 157 patients who have been treated in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one prescription for Lorcaserin treatment
* At least 18 years of age or with guardian/parent able to consent for a minor

Exclusion Criteria:

- Patient under the age of 18 at time of index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population includes 157 patients seen and evaluated in an insurance-based medical weight loss clinic in San Diego, CA. Eligible participants will include patients who are overweight or obese, and who received at least one prescription for Lorcaserin treatment.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Weight change - in pounds | Up to 1 year of medication use
  Change in weight with Lorcaserin treatment
Duration of Use - in weeks | Up to 1 year of medication use
  Average duration of treatment with Lorcaserin

SECONDARY OUTCOMES:
Change in heart rate | Up to 1 year of medication use
  Assessment of change heart rate (bpm)
Change in blood pressure | Up to 1 year of medication use
  Assessment of change in both systolic and diastolic blood pressure (mmHg)
Change in lipid levels | Up to 1 year of medication use
  Assessment of change in lab values for total cholesterol, LDL, HDL and Triglycerides
Change in liver enzymes | Up to 1 year of medication use
  Assessment of change in lab values for AST and ALT
Change in glucose values | Up to 1 year of medication use
  Assessment of change in lab values for fasting glucose and hemoglobin A1c

OTHER OUTCOMES:
Reasons for Discontinuation | Up to 1 year of medication use
  Reasons for discontinuing treatment with Lorcaserin - as obtained by annotation in patient's medical record from overseeing physician.
Changes in Healthcare Utilization | Up to 1 year of medication use
  Assessment of changes in healthcare utilization including all Scripps outpatient medical visits, visits to the ER and/or Urgent care, and inpatient hospitalizations. All of the above are assessed via the Scripps network EMR and only include visits made to a Scripps facility. Reason for visit and level of visit billed reviewed via EMR using billing and diagnosis codes.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Fujioka, MD, Principal Investigator — Scripps Clinic Medical Group
Locations (1):
- Scripps Whittier Diabetes Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No